CLINICAL TRIAL: NCT06718036
Title: Validation and Evaluation of the ICF Rehabilitation Set: a Polish Clinical Perspective
Brief Title: Validation and Evaluation of the ICF Rehabilitation Set
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Agnieszka Wiśniowska-Szurlej, PhD, University of Rzeszow
Other Study IDs: ICF Rehabilitation Set
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Disease
Keywords: Disability; Rehabilitation; ICF
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults participating in the therapeutic rehabilitation process
  Interventions: Other: Validation and evaluation of the use of the ICF Rehabilitation Set in clinical practice

INTERVENTIONS:
Other: Validation and evaluation of the use of the ICF Rehabilitation Set in clinical practice — Validation and evaluation of the use of the ICF Rehabilitation Set in clinical practice

SUMMARY:
Rehabilitation is considered a key health strategy in the 21st century. The aim of rehabilitation is to optimize the functioning of patients. The International Classification of Functioning, Disability and Health (ICF) is a framework for describing and organizing information on functioning and disability. Therefore, the aim of the study is to validate and evaluate the application of the ICF Rehabilitation Set in Polish clinical practice.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO) rehabilitation is defined as "a set of interventions designed to optimize functioning and reduce disability in individuals with health conditions in interaction with their environment." Rehabilitation is considered a key health strategy in the 21st century. Demographic and epidemiological trends indicate that human functioning is one of the most important indicators of population health, apart from morbidity and mortality. Thus, it suggests that the main focus of healthcare will be on the real health needs generated by long-term treatment of chronic diseases, including comprehensive enhancement and intensification of rehabilitation.

The aim of rehabilitation is to optimize functioning of patients. WHO indicates International Classifications and Terminologies including the International Statistical Classification of Diseases and Related Health Problems (ICD) and the International Classification of Functioning, Disability and Health (ICF) as the global standards for collecting data regarding health, clinical documentation and statistical data aggregation3. ICF and ICD provide health information in relation to diagnosis (ICD) as well as functioning and disability (ICF). The ICF is based on a holistic biopsychosocial disability model that allows for a comprehensive and wide approach to the problems of an individual related to functioning in his/her living environment.

A Polish version of the ICF Rehabilitation Set has been developed, which contains 29 categories and is proposed as framework for harmonizing information on the functioning and disability of people participating in the rehabilitation process. Therefore, the aim of the study is to validate and assess the use of the ICF Rehabilitation Set in Polish clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic diseases, including: neurological, cardiological, pulmonary and musculoskeletal problems.
* Cognitive state, enabling to answer questions reliably and accurately, minimum 6 points on the AMTS scale
* Adults participating in the rehabilitation process
* Consent to participate in the study.

Exclusion Criteria:

* Previous surgeries, with surgical intervention.
* Fractures.
* Severe systemic diseases that prevent the examination, e.g. acute neoplastic disease, exacerbation of chronic diseases, infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults participating in the therapeutic rehabilitation process
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
ICF Rehabilitation Set | Time Frame: 2024-12/2025-06]

SECONDARY OUTCOMES:
Index Barthel | Time Frame: 2024-12/2025-06]

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rzeszow, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wisniowska-Szurlej A, Sozanska A, Brozonowicz J, Wilmowska-Pietruszynska A, Sozanski B. Validation and evaluation of the application of the ICF Rehabilitation Set: a Polish clinical perspective. BMC Health Serv Res. 2025 Aug 5;25(1):1027. doi: 10.1186/s12913-025-13048-2. PMID 40764554